CLINICAL TRIAL: NCT06332846
Title: Assessment of Oral Health in Patients Hospitalized Because of Ischemic Stroke
Brief Title: Oral Health in Patients Hospitalized Because of Ischemic Stroke
Status: Completed | Type: Observational
Sponsor: Pomeranian Medical University Szczecin (Other)
Responsible Party: Sponsor
Other Study IDs: KB-0012/06/10
Record Dates: First submitted 2024-03-01; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Oral Disease; Stroke, Ischemic
Keywords: stroke; oral health; dentition; periodontium
MeSH Terms: conditions — Mouth Diseases; Ischemic Stroke; Stroke | interventions — Diagnosis, Oral; Control Groups

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: The study group consisted of 59 individuals subjects with a first ischemic stroke, with symptoms from the anterior cerebral artery (basin of the internal carotid artery), with a significant neurological deficit (minimum 3 points according to National Institute of Health Stroke Scale
  Interventions: Other: oral examination
- control group: The control group (59 individuals) matched for age and gender was selected among patients of the Department of Interdisciplinary Dentistry at Pomeranian Medical University in Szczecin.
  Interventions: Other: oral examination

INTERVENTIONS:
Other: oral examination — The oral health was assessed in each patient enrolled in the study. The examination was performed by using dental mirror and a calibrated periodontal probe in a day ight
  Other Names: study group
  Groups: control group
Other: oral examination — The oral health was assessed in each patient enrolled in the study. The examination was performed by using dental mirror and a calibrated periodontal probe in the artificial lightning
  Other Names: control group
  Groups: study group

SUMMARY:
Maintaining good oral health is essential for general health and quality of life. Results of many anal-yses showed that stroke patients had poorer oral condition and worse periodontal status than control population. The aim of the study was to carry out a clinical observation concerning condition of oral health in stroke patients and healthy population.

The oral health was assessed in patients with stroke and in (control group). The following elements were assessed: missing teeth, the presence of active caries foci, the presence of existing fillings and prosthetic restorations. To assess oral hygiene API (Approximal Plaque Index) was used. As part of periodontal examina-tion, the following were assessed: the presence of dental deposits, the depth of the existing periodontal pockets, tooth mobility according to Hall and Sulcus Bleeding Index during probing (SBI).

ELIGIBILITY:
Inclusion Criteria:

* first ischemic stroke, with symptoms from the anterior cerebral artery (basin of the internal carotid artery), with a significant neurological deficit (minimum 3 points according to National Institute of Health Stroke Scale (NIHSS))

Exclusion Criteria:

* aphasia, disturbances of consciousness, mental disorders- making it impossible to express informed consent,
* surgery of the salivary glands- disrupting the secretion of saliva,
* diseases that disrupt salivary secretion (diabetes mellitus, Sjogren's syndrome, condition after radio-therapy in the area of the salivary glands)

Ages: 45 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study group consisted of 59 individuals subjects with a first ischemic stroke, with symptoms from the anterior cerebral artery (basin of the internal carotid artery), with a significant neurological deficit (minimum 3 points according to National Institute of Health Stroke Scale (NIHSS)). The control group (59 individuals) matched for age and gender was selected among patients of the Department of Interdisciplinary Dentistry at Pomeranian Medical University in Szczecin.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
Oral health status | Baseline
  The study aimed to estimate and compare a condition of oral health in stroke patients during hospital stay and healthy individuals.The following elements were assessed: a number of missing teeth, active caries foci and existing fillings. Each tooth was evaluated and scored as sound, decayed (DT), extracted because of the carious pro-cess (MT), or filled due to caries (FT). The data obtained from the examination were used to calculate the DMFT index, which is the sum of DT, MT and FT, and expresses dental caries experience.
Oral hygiene assessment | Baseline
  Value of API is determined in percentage, according to proportion of the number of interproximal areas with plaque to number of all assessed interproximal areas.API values between 100-70% indicate the improper oral hygiene, values between 70-40% indicate an average oral hygiene, values between 39-25% indicate quite good hygiene, and values below 25% indicate optimal oral hygiene.
Periodontal status- periodontal pockets | Baseline
  The depth of the existing periodontal pockets in mm (up to 3mm, 3-6 mm, above 6 mm).
Periodontal status-tooth mobility | Baseline
  Tooth mobility according to Hall (0- no mobility, 1- labio-lingual mobility up to 1mm, 2- labio-lingual mobility up to 2 mm, 3- labio-lingual and vertical mobility).
Periodontal status- bleeding | Baseline
  Sulcus Bleeding Index during probing (SBI). SBI is an index of gingival inflammation in which bleeding is measured from four gingival units (mesial and distal papillary units and labial and lingual marginal units) using a periodontal probe with a 0,5 mm diameter tip. The scoring range around eight anterior teeth (four maxillary and four mandibular) is from 0 (healthy appearance and no bleeding on probing to 5 (spontaneous bleeding with marked swelling and change in colour).

CONTACTS AND LOCATIONS:
Locations (1):
- Pomeranian Medical University in Szczecin, Szczecin, Poland